CLINICAL TRIAL: NCT02928692
Title: Minocycline Attenuate Postoperative Cognitive Dysfunction and Delirium: A Multicenter, Randomized, Double-Blind Clinical Trail
Brief Title: Minocycline Attenuate Postoperative Cognitive Dysfunction and Delirium
Acronym: MAPOCD
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: RenJi Hospital (Other)
Collaborators: Shanghai 10th People's Hospital (Other); Pudong New Area People's Hospital (Unknown); Shanghai Pudong Hospital (Other); Shanghai Pudong New Aera Dongming Community Health Care Center (Unknown)
Responsible Party: Principal Investigator, diansan su, Dr., RenJi Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 20158202
Record Dates: First submitted 2016-10-05; First posted 2016-10-10 (Estimated); Last update posted 2020-01-28 (Actual); Status verified 2020-01

CONDITIONS: Prostate Cancer; Carcinoma of the Rectum; Colon Cancer; Renal Carcinoma
Keywords: Minocycline; Postoperative cognitive dysfunction; Postoperative delirium
MeSH Terms: conditions — Prostatic Neoplasms; Rectal Neoplasms; Colonic Neoplasms; Carcinoma, Renal Cell; cyclopia sequence; Postoperative Cognitive Complications; Emergence Delirium | interventions — Minocycline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- Placebo (Placebo Comparator): Placebo administered before surgery
  Interventions: Drug: Placebo
- Minocycline (Experimental): Minocycline was administrated before surgery
  Interventions: Drug: Minocycline
- Volunteers (No Intervention): Health people for calculate the incidence of POCD

INTERVENTIONS:
Drug: Minocycline
  Arms: Minocycline
Drug: Placebo
  Arms: Placebo

SUMMARY:
Postoperative cognitive dysfunction (POCD) and postoperative delirium occurs mainly in aged patients. POCD and POD may increase the mortality and morbidity. However, the mechanism of POCD is not clear yet and no effective therapy method was proved. According to previous study, the neuroinflammation is the main reason both for POCD and POD. Minocycline is a tetracycline derivative. Due to it's lipophilic structure, it is easy to pass through blood brain barrier and attenuate neuroinflammation. It's neuroprotective effects has been proven in many experimental animal models such as Alzheimer's disease, Huntington's disease and Parkinson's syndrome. In present study, the investigators hypothesized that minocycline would attenuate the incidence of POCD and POD in the aged patients.

ELIGIBILITY:
For the placebo and minocycline group;

Inclusion Criteria:

1. Elder than 65 years old
2. Speak Chinese Mandarin
3. Those who will undergo major general surgery like colorectal cancer excision, major urinary surgery like radical prostatectomy and radical nephrectomy
4. Signed the inform consent
5. American Society of Anesthesiologists classification I to III

Exclusion Criteria:

1. Existing cerebral disease, or have a history of neurological and psychiatric diseases including Alzheimer Disease, stroke, epilepsy and psychosis;
2. Existing cognitive impairment as evidenced by Mini-Mental State Examination scores below 24;
3. Severe audition or vision disorder;
4. Unwillingness to comply with the protocol or procedures.
5. Cannot communicated with Chinese Mandarin
6. With severe skin disease
7. Serious heart or liver or renal insufficiency patients
8. Had surgery in the past 30 days
9. Allergy to tetracycline or minocycline

For the health volunteers;

Inclusion Criteria:

1. Elder than 65 years old
2. Speak Chinese Mandarin
3. Signed the inform consent
4. No major disease health people

Exclusion Criteria:

1. Existing cerebral disease, or have a history of neurological and psychiatric diseases including Alzheimer Disease, stroke, epilepsy and psychosis;
2. Existing cognitive impairment as evidenced by Mini-Mental State Examination scores below 24;
3. Severe audition or vision disorder;
4. Unwillingness to comply with the protocol or procedures.
5. Cannot communicated with Chinese Mandarin
6. Drug abuse, alcoholism
7. Serious heart or liver or renal insufficiency patients
8. Had surgery in the past 30 days
9. Plan to undergo surgery in the following 3 months.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 750 (Estimated)
Dates: Start 2016-11 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
POCD incidence 7 days (or before leaving hospital) after surgery | 7 days (or before leaving hospital)
POD incidence | 1 to 5 days after surgery

SECONDARY OUTCOMES:
POCD incidence 2 months after surgery | 2 months after surgery

CONTACTS AND LOCATIONS:
Locations (5):
- China (5):
  - Scales, Shanghai, Shanghai Municipality
  - Shanghai Pudong Hospital, Shanghai
  - Shanghai Pudong New Area Dongming Community Health Care Center, Shanghai
  - Shanghai Pudong New Area people's Hopsital, Shanghai
  - Shanghai Tenth Hospital, Shanghai

REFERENCES:
- [Background] Large MC, Reichard C, Williams JT, Chang C, Prasad S, Leung Y, DuBeau C, Bales GT, Steinberg GD. Incidence, risk factors, and complications of postoperative delirium in elderly patients undergoing radical cystectomy. Urology. 2013 Jan;81(1):123-8. doi: 10.1016/j.urology.2012.07.086. Epub 2012 Nov 13. PMID 23153950
- [Background] Pol RA, van Leeuwen BL, Izaks GJ, Reijnen MM, Visser L, Tielliu IF, Zeebregts CJ. C-reactive protein predicts postoperative delirium following vascular surgery. Ann Vasc Surg. 2014 Nov;28(8):1923-30. doi: 10.1016/j.avsg.2014.07.004. Epub 2014 Jul 10. PMID 25017770
- [Background] Nadelson MR, Sanders RD, Avidan MS. Perioperative cognitive trajectory in adults. Br J Anaesth. 2014 Mar;112(3):440-51. doi: 10.1093/bja/aet420. Epub 2014 Jan 2. PMID 24384981
- [Background] Westhoff D, Witlox J, Koenderman L, Kalisvaart KJ, de Jonghe JF, van Stijn MF, Houdijk AP, Hoogland IC, Maclullich AM, van Westerloo DJ, van de Beek D, Eikelenboom P, van Gool WA. Preoperative cerebrospinal fluid cytokine levels and the risk of postoperative delirium in elderly hip fracture patients. J Neuroinflammation. 2013 Oct 7;10:122. doi: 10.1186/1742-2094-10-122. PMID 24093540
- [Background] Shim JJ, Leung JM. An update on delirium in the postoperative setting: prevention, diagnosis and management. Best Pract Res Clin Anaesthesiol. 2012 Sep;26(3):327-43. doi: 10.1016/j.bpa.2012.08.003. PMID 23040284
- [Background] van Meenen LC, van Meenen DM, de Rooij SE, ter Riet G. Risk prediction models for postoperative delirium: a systematic review and meta-analysis. J Am Geriatr Soc. 2014 Dec;62(12):2383-90. doi: 10.1111/jgs.13138. PMID 25516034
- [Background] American Geriatrics Society Expert Panel on Postoperative Delirium in Older Adults. Postoperative delirium in older adults: best practice statement from the American Geriatrics Society. J Am Coll Surg. 2015 Feb;220(2):136-48.e1. doi: 10.1016/j.jamcollsurg.2014.10.019. Epub 2014 Nov 14. No abstract available. PMID 25535170
- [Background] Bellelli G, Mazzola P, Morandi A, Bruni A, Carnevali L, Corsi M, Zatti G, Zambon A, Corrao G, Olofsson B, Gustafson Y, Annoni G. Duration of postoperative delirium is an independent predictor of 6-month mortality in older adults after hip fracture. J Am Geriatr Soc. 2014 Jul;62(7):1335-40. doi: 10.1111/jgs.12885. Epub 2014 Jun 2. PMID 24890941
- [Background] Ramaiah R, Lam AM. Postoperative cognitive dysfunction in the elderly. Anesthesiol Clin. 2009 Sep;27(3):485-96, table of contents. doi: 10.1016/j.anclin.2009.07.011. PMID 19825488
- [Background] Sauer AM, Kalkman C, van Dijk D. Postoperative cognitive decline. J Anesth. 2009;23(2):256-9. doi: 10.1007/s00540-009-0744-5. Epub 2009 May 15. PMID 19444566
- [Background] Moller JT, Cluitmans P, Rasmussen LS, Houx P, Rasmussen H, Canet J, Rabbitt P, Jolles J, Larsen K, Hanning CD, Langeron O, Johnson T, Lauven PM, Kristensen PA, Biedler A, van Beem H, Fraidakis O, Silverstein JH, Beneken JE, Gravenstein JS. Long-term postoperative cognitive dysfunction in the elderly ISPOCD1 study. ISPOCD investigators. International Study of Post-Operative Cognitive Dysfunction. Lancet. 1998 Mar 21;351(9106):857-61. doi: 10.1016/s0140-6736(97)07382-0. PMID 9525362
- [Background] Monk TG, Weldon BC, Garvan CW, Dede DE, van der Aa MT, Heilman KM, Gravenstein JS. Predictors of cognitive dysfunction after major noncardiac surgery. Anesthesiology. 2008 Jan;108(1):18-30. doi: 10.1097/01.anes.0000296071.19434.1e. PMID 18156878
- [Background] Steinmetz J, Christensen KB, Lund T, Lohse N, Rasmussen LS; ISPOCD Group. Long-term consequences of postoperative cognitive dysfunction. Anesthesiology. 2009 Mar;110(3):548-55. doi: 10.1097/ALN.0b013e318195b569. PMID 19225398
- [Background] Vacas S, Degos V, Feng X, Maze M. The neuroinflammatory response of postoperative cognitive decline. Br Med Bull. 2013;106(1):161-78. doi: 10.1093/bmb/ldt006. Epub 2013 Apr 4. PMID 23558082
- [Background] Wan Y, Xu J, Ma D, Zeng Y, Cibelli M, Maze M. Postoperative impairment of cognitive function in rats: a possible role for cytokine-mediated inflammation in the hippocampus. Anesthesiology. 2007 Mar;106(3):436-43. doi: 10.1097/00000542-200703000-00007. PMID 17325501
- [Background] Fidalgo AR, Cibelli M, White JP, Nagy I, Maze M, Ma D. Systemic inflammation enhances surgery-induced cognitive dysfunction in mice. Neurosci Lett. 2011 Jul 1;498(1):63-6. doi: 10.1016/j.neulet.2011.04.063. Epub 2011 May 6. PMID 21575676
- [Background] Cibelli M, Fidalgo AR, Terrando N, Ma D, Monaco C, Feldmann M, Takata M, Lever IJ, Nanchahal J, Fanselow MS, Maze M. Role of interleukin-1beta in postoperative cognitive dysfunction. Ann Neurol. 2010 Sep;68(3):360-8. doi: 10.1002/ana.22082. PMID 20818791
- [Background] Terrando N, Eriksson LI, Ryu JK, Yang T, Monaco C, Feldmann M, Jonsson Fagerlund M, Charo IF, Akassoglou K, Maze M. Resolving postoperative neuroinflammation and cognitive decline. Ann Neurol. 2011 Dec;70(6):986-995. doi: 10.1002/ana.22664. PMID 22190370
- [Background] Vacas S, Degos V, Tracey KJ, Maze M. High-mobility group box 1 protein initiates postoperative cognitive decline by engaging bone marrow-derived macrophages. Anesthesiology. 2014 May;120(5):1160-7. doi: 10.1097/ALN.0000000000000045. PMID 24162463
- [Background] Wan Y, Xu J, Meng F, Bao Y, Ge Y, Lobo N, Vizcaychipi MP, Zhang D, Gentleman SM, Maze M, Ma D. Cognitive decline following major surgery is associated with gliosis, beta-amyloid accumulation, and tau phosphorylation in old mice. Crit Care Med. 2010 Nov;38(11):2190-8. doi: 10.1097/CCM.0b013e3181f17bcb. PMID 20711073
- [Background] Su X, Feng X, Terrando N, Yan Y, Chawla A, Koch LG, Britton SL, Matthay MA, Maze M. Dysfunction of inflammation-resolving pathways is associated with exaggerated postoperative cognitive decline in a rat model of the metabolic syndrome. Mol Med. 2013 Feb 8;18(1):1481-90. doi: 10.2119/molmed.2012.00351. PMID 23296426